CLINICAL TRIAL: NCT06803186
Title: Effect of High Power Laser Therapy on Myoelectrical Activities of Suboccipital Muscles and Quality of Life in Patients With Cervicogenic Headache
Brief Title: High Power Laser on Suboccipital Myoelectrical Activities and Quality of Life in Patients With Cervicogenic Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Karem Youssef Tawfik, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005470
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power laser therapy and conventional physical therapy program (Experimental): The participants will receive high power laser therapy (HPLT) for 15 minutes in addition to a conventional physical therapy program (therapeutic exercise) for 45 minutes three a week for six weeks.
  Interventions: Device: High-power laser therapy; Other: Conventional physical therapy program
- Placebo high power laser therapy and conventional physical therapy program (Active Comparator): The participants will receive placebo high power laser therapy (HPLT) for 15 minutes in addition to a conventional physical therapy program (therapeutic exercise) for 45 minutes three a week for six weeks.
  Interventions: Device: Placebo (PL) high power laser; Other: Conventional physical therapy program

INTERVENTIONS:
Device: High-power laser therapy — High power laser therapy (HPLT) with a neodymium-yttrium aluminum garnet laser with a pulsating waveform produced by a ( Hilterapia device , ASA, Arcugnano, Vicenza, Italy). It will be set at the following parameters: Nd:YAG laser with pulsed emission (1064 nm), very high peak powers with average power 6 W, high levels of fluency (760 mJ/cm energy density), short pulse duration (250 μs), low frequency (10-40 Hz), and 5-cm probe diameter for 15 minutes.
  The scanning will be performed longitudinally &transversely from the C3 to C7 posterior neck in the paraspinal region, upper back, inter-scapular area, trapezius, sternocleidomastoid muscles, and posterior & lateral shoulder areas
  Arms: High power laser therapy and conventional physical therapy program
Device: Placebo (PL) high power laser — laser probe scanning will be applied to the same areas as that applied in the HPLT procedure. PL will be applied while the lights of the device will be on, with no current flowing through the device. Placebo therapy will be applied at the same frequency as HPLT (Three sessions a week for six weeks for a total of 18 sessions; one session will be lasted 15 minutes).
  Arms: Placebo high power laser therapy and conventional physical therapy program
Other: Conventional physical therapy program — A specific program of 45-min exercise of three sessions a week for six weeks for a total of 18 sessions. Corrective exercises will be performed initially by stretching exercises for(suboccipital, upper trapezeius, scalene, levator scapulae, sternocleidomastoid, pectoralis major/minor muscles) will be given four repetitions with 30 second hold. each with 3 seconds rest between each stretch Then, strengthening exercises will be performed initially in an isometric manner for weak muscles (deep cervical flexors, rhomboidus, and lower trapezeius muscles) will be done initially without weight and afterward by using Theraband and dumbells. All patients will be instructed to achieve three sets of 12 repetitions of the strengthening exercises (isometrics exercises) with 1 to 2 minutes rest in between each set. Contraction will be held for 5 seconds/repetitions. 10-20 repetitions for strengthening exercises and 3 sets of 30 repetitions for endurance exercise

SUMMARY:
The study will be conducted:

To investigate the effect of high-power laser on myoelectrical activities of suboccipital muscles in patients with cervicogenic headache.

* To investigate the effect of high-power laser on pain in patients with cervicogenic headache.
* To investigate the effect of high-power laser on quality of life in patients with cervicogenic headache.

DETAILED DESCRIPTION:
Cervicogenic headache is a classification of headache in which pain is referred from the cervical spine. This category of headache is typically chronic, presented as unilateral cephalgia, spreading over the occipital, temporal, and frontal regions and is believed to be caused by musculoskeletal dysfunction of the neck.

In high-power laser therapy (HPLT) there is an increase in mitochondrial oxidative reaction and adenosine phosphate (photobiology effect). The pain-releasing effect of HPLT is provided by reducing the transmission of painful stimuli and increased morphine mimetic factors. It has rapidly induced photochemical and photothermal effects, increasing blood flow, cell metabolism, and vascular permeability.

In a recent study on exercise for cervicogenic headache, Subjects reported significant decreases in the frequency, intensity, and duration of their headaches.

To our knowledge there is no study was found to investigate the effect of high-power laser therapy (HPLT) on myoelectrical activities of suboccipital muscles, pain and functional activities in patients with cervicogenic headache.

So, this study aimed to determine the effect of high power laser therapy (HPLT) on myoelectrical activities of suboccipital muscles , pain and quality of life in patients with cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from cervicogenic headache based on international headache society "IHS" criteria for cervicogenic headache.
* Unilateral cervical radiculopathy (Upper cervical C1 -C4).
* Age ranged from 30 to 50 years.
* Neck pain referring unilaterally to suboccipital region.
* The pain and restriction in C1-C2 rotation by Cervical Flexion-Rotation Test (FRT )
* Intensifying headache by manual pressure to upper cervical muscles and joints.
* Experiencing headache at least once per week for the last 6 months.
* Patients will be referred by neurological consultants.
* Body mass index (18.5 - 29. 9 Kg/m2).
* Moderate (45-74) to severe (75-100) neck pain on the visual analogue scale.

Exclusion Criteria:

* Cervical myelopathy, cervical instability, cervical fracture cervical surgery with evidence of pyramidal, posterior column disorders.
* History of any neurologic disease ( stroke, MS , cerebellar disorders , vestibular dysfunction and neuropathy )Pregnant or breastfeeding women
* Other types of headaches (migraine - cluster headaches- tension headache)
* Patients of systemic diseases such as rheumatoid arthritis
* contraindication to high-power Laser such as:
* Wounds or skin changes in the neck or shoulder region (such as psoriasis, scars, or burns).
* Photosensitivity diagnosis.
* Tumors of some type have been diagnosed in the last 5 years.
* Presence of solar urticaria or adverse reactions to sunlight.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Myoelectrical activity of suboccipital muscle | 6 weeks
  Needle electromyography (EMG, Micromed, made in Italy) is a definitive invasive technique that allows an objective evaluation of muscle activity.
  Activation pattern of the suboccipital muscle mainly the rectus capitis posterior muscles will be recorded and analyzed. The skin is cleaned with alcohol to reduce skin impedance. A Concentric needle is inserted in the rectus capitis posterior muscles, positioned caudad, at a point 1-2cm lateral to the midline at the level of the approximation of the posterior arch of C1. at approximately 80 degrees from an imaginary line drawn parallel to the surface of the skin in the mid-sagital plane. The patient performed extension delivering maximum voluntary contraction against therapist hand. Reference electrode is placed just above the middle of the spine of the right scapula or over the forehead. Data will be represented as interference patterns (graphics), analyzed and compared before and after the intervention for all participants in the study.
Neck Disability Index (NDI) | 6 weeks
  The NDI will be used to assess neck pain and quality of life for all participants before and after the treatment program. It is consisted of 10 items with six potential responses per item relating to pain severity, headache, attention, and various physical activities (lifting, personal care, recreation, work, driving, reading, and sleeping). Each item's score ranges from 0 to 5. The maximum possible total score is 50, which is translated to a percentage. Higher scores indicate a greater degree of impairment. The NDI has been demonstrated to be a valid, had stable psychometric characteristics and accurate questionnaire for people suffering from neck pain
Quality of life (QoL) assessment | 6 weeks
  The SF-36 questionnaire will be used to assess QoL for all participants before and after the end of the study program. It is a self-administered questionnaire containing 36 items which takes about five minutes to complete. It measures health on eight multi-item dimensions, covering physical functioning, role limitation due to physical health, bodily pain, general health perception, vitality, social functioning, role limitation due to emotional problems and perceived mental health. Each domain contains number of items. The answers to each question are extrapolated to a standardized set of answers, and the results are transferred to a scale of 0-100, where 0 represents the worst state of health measured, and 100 represents the best state of health measured. It has good validity and reliability and can be used as a general questionnaire to assess quality of life.

SECONDARY OUTCOMES:
Pain intensity | 6 weeks
  Visual analogue scale (VAS) will be used to assess pain intensity for all participants before and after the treatment program. It is a straight line, and its length is 10 cm, ranging from no pain or discomfort (zero), to the worst pain (10) that the patient could feel. it is a valid scale and has good validity and reliability.
Headache impact test-6 (The HIT-6) | 6 weeks
  The six-item Headache Impact Test (HIT-6) from Quality Metric is a patient-reported outcome (PRO) tool used to capture the impact of headaches and headache treatments on functional health and wellbeing. The HIT-6 addresses six core domains affected by headaches: pain. social Functioning, role Functioning, cognitive Functioning, vitality and psychological Stress.
  Each item is answered on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The final score is obtained from a simple summation of the six items. The HIT-6 total score ranges between 36 and 78, with larger scores reflecting greater impact. Four categories have been derived to aid in the interpretation of HIT-6 scores: scores ≤49 represent little or no impact; scores between 50 and 55 represent mild impact; scores between 56 and 59 represent moderate impact; and scores ≥60 indicate severe impact.

CONTACTS AND LOCATIONS:
Overall Officials: Shehab Khadrawy, Professor, Study Director — Al-Azhar University; Asharaf A. Abdelmoneim, Professor, Study Director — Cairo University; Abd El-Aleem A Attia, professor, Study Chair — Cairo University
Locations (1):
- Ahmed Karem Youssef Tawfik, Cairo, Egypt